CLINICAL TRIAL: NCT06845800
Title: Microneurography and Microneurostimulation for Prognosis and Rehabilitation of Disorders of Consciousness
Brief Title: Peripheral Nerve Stimulation for Prognostic and Diagnostic Biomarker Identification in Disorders of Consciousness
Acronym: MICRO-DOC
Status: Completed | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Scuola Superiore Sant'Anna Pisa (Unknown)
Responsible Party: Sponsor
Other Study IDs: TUNEBEAM_MICRODOC
Record Dates: First submitted 2025-02-17; First posted 2025-02-25 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-02

CONDITIONS: Disorders of Consciousness Due to Severe Brain Injury
Keywords: Electroencephalography; Near-Nerve Stimulation; Prognosis; Diagnosis; Neurorehabilitation; Disorder of Consciousness
MeSH Terms: conditions — Disease; Consciousness Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Disorders of Consciousness admitted to the Intensive Rehabilitation Unit: Patients admitted with a Disorder of Consciousness to the Intensive Rehabilitation Unit (IRU) of Fondazione Don Carlo Gnocchi (Florence).
  * Age ≥ 18 years, both sexes;
  * Severe Acquired Brain Injury (ABI), regardless of etiology;
  * Patients with a severe alteration of consciousness due to severe ABI of various etiologies, including Cardiac Arrest, Traumatic Brain Injury, Cerebral Ischemia, or Hemorrhage;
  * Signed informed consent provided by a family member, caregiver, or legal guardian.

SUMMARY:
This observational study aims to integrate anamnestic, clinical, and innovative neurophysiological data to assess their impact on the diagnosis and prognosis of patients with Disorders of Consciousness. The main questions it aims to answer are:

* Is it possible to identify biomarkers with high diagnostic relevance for distinguishing subcategories of patients with Disorders of Consciousness?
* Can biomarkers with potential medium- and long-term prognostic value be identified for each category of patients with Disorders of Consciousness?

Participants will undergo an EEG examination during near-nerve stimulation of the median nerve. Clinical and anamnestic data will also be recorded and collected at follow-up.

DETAILED DESCRIPTION:
At the enrollment of each patient with Disorders of Consciousness, demographic, anamnestic, and clinical data are prospectively collected. The etiology is categorized as traumatic, anoxic, hemorrhagic, or ischemic. The lesion side is defined according to the latest CT scans from the acute phase and is grouped as left, right, and bilateral. All patients undergo a standard neurophysiological evaluation, and the level of consciousness is assessed using the CRS-R scale following international guidelines. It is repeated to confirm the clinical status of the patient, and a reduction of sedation is performed if deemed safe by the physician. Two months after admission to the IRU, the neurophysiological and consciousness assessments are repeated.

In addition to clinical and standard neurophysiological evaluations, two types of SSEPs are acquired during continuous EEG recording through both Surface Cutaneous Stimulation (SCS) and Near-Nerve Stimulation (NNS) of the median nerve. EEG signals are collected using a 61-channel cap with a sampling rate of 512 Hz.

The electrical stimulation is applied over the median nerve proximally to the wrist, and the stimulation side is chosen contralaterally to the less affected hemisphere. Superficial bipolar electrodes are used for SCS, whereas a microneedle with 1 MΩ of impedance is inserted under the skin for NNS. The electrical pulse of 0.2 ms is delivered at a rate of 1 Hz in two sets of 50 repetitions. The stimulation amplitude is chosen as the minimum value able to generate a response only in sensory or sensory-motor fibers for NNS and SCS, respectively. The only sensory activation in NNS is preferred to minimize the influence of motor twitches on brain responses. For SCS, due to the difficulty of exclusively stimulating sensory fibers, the amplitude is set as the minimal value required to elicit both sensory and motor activation.

To monitor the stimulated fibers, the peripheral pathway of the median nerve is recorded. In particular, surface electrodes are positioned on the three fingers innervated by the median nerve for the acquisition of Sensory Nerve Action Potential (SNAP) and on the palm proximally to the motor twitch for the acquisition of Compound Motor Action Potential (CMAP). This information is essential in patients with DoC for different reasons:

i) Identifying the proximity to the median nerve, a crucial step due to the unresponsiveness and lack of cooperation of this population.ii) Identifying the type of active fibers.iii) Monitoring feedback to confirm the accurate placement of the microelectrode.

Whenever the minimum amplitude evokes a CMAP/SNAP, the related amplitude is selected for SCS/NNS. The device automatically extracts the mean values of amplitude and latency of CMAP/SNAP during the experimental session.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years, both sexes;
* Severe acquired brain injury (regardless of etiology);
* Patients with severe alteration of consciousness state due to severe acquired brain injury of various etiologies (Cardiac Arrest, Traumatic Brain Injury, Cerebral Ischemia or Hemorrhage);
* Informed consent signature by family member/caregiver/legal guardian.

Exclusion Criteria:

* Time since the acute event greater than 3 months;
* Previous neurological diseases;
* Previous acute brain injuries, psychiatric disorders, neurodegenerative diseases, neoplasms, severe systemic diseases;
* Modified Barthel Index pre-event < 50;
* Unstable medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were admitted with a Disorder of Consciousness to the Intensive Rehabilitation Unit (IRU) of Fondazione Don Carlo Gnocchi (Florence).
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Identification of Neurophysiological Diagnostic Biomarkers in Disorders of Consciousness | From enrollment to the baseline experimental session (within 7 days from enrollment)
  Quantification of the Agreement Between Newly Proposed Neurophysiological Markers From Near-Nerve Stimulation Examinations and Disorders of Consciousness Classification Based on the Coma Recovery Scale-Revised (UWS, MCS-, MCS+)
Identification of Neurophysiological Prognostic Biomarkers in Disorders of Consciousness | From enrollment to the end of follow up at 6-months from baseline assessment
  Quantification of Prognostic Prediction Accuracy of Newly Proposed Neurophysiological Markers From Near-Nerve Stimulation in Classifying Disorders of Consciousness Based on the Coma Recovery Scale - Revised (UWS, MCS-, MCS+, EMCS)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi, Florence, FI, Italy

IPD SHARING:
Plan to Share IPD: Yes
Upon publication of results, anonymized data and analysis code will be shared to ensure reproducibility. Zenodo and GitHub repositories will be created.
Supporting Information: SAP, Analytic Code
Time Frame: Upon publication of results
Access Criteria: Data and code will be available for research purposes upon request to authors.

REFERENCES:
- [Background] Vallbo AB. Microneurography: how it started and how it works. J Neurophysiol. 2018 Sep 1;120(3):1415-1427. doi: 10.1152/jn.00933.2017. Epub 2018 Jun 20. PMID 29924706
- [Background] Mano T, Iwase S, Toma S. Microneurography as a tool in clinical neurophysiology to investigate peripheral neural traffic in humans. Clin Neurophysiol. 2006 Nov;117(11):2357-84. doi: 10.1016/j.clinph.2006.06.002. Epub 2006 Aug 10. PMID 16904937
- [Background] Hakiki B, Donnini I, Romoli AM, Draghi F, Maccanti D, Grippo A, Scarpino M, Maiorelli A, Sterpu R, Atzori T, Mannini A, Campagnini S, Bagnoli S, Ingannato A, Nacmias B, De Bellis F, Estraneo A, Carli V, Pasqualone E, Comanducci A, Navarro J, Carrozza MC, Macchi C, Cecchi F. Clinical, Neurophysiological, and Genetic Predictors of Recovery in Patients With Severe Acquired Brain Injuries (PRABI): A Study Protocol for a Longitudinal Observational Study. Front Neurol. 2022 Feb 28;13:711312. doi: 10.3389/fneur.2022.711312. eCollection 2022. PMID 35295839